CLINICAL TRIAL: NCT04521660
Title: The Effect of Using Virtual Reality Glasses on Pain, Anxiety and Hemodynamic Parameters During Coronary Angiography: A Randomized Controlled Trial
Brief Title: The Effect of Using Virtual Reality Glasses During Coronary Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, PhD, Asst Prof, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-94
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-02

CONDITIONS: Coronary Angiography
Keywords: virtual reality; pain; anxiety; hemodynamic parameters; angiography
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will wear virtual reality glasses during coronary angiography.
  Interventions: Device: Virtual reality glasses
- Control group (No Intervention): Patients in the control group will not wear virtual reality glasses. They will be given standard care and treatment during the procedure.

INTERVENTIONS:
Device: Virtual reality glasses — Virtual reality (VR) is a new method that can be used to distract and prepare patients for the procedure during medical procedures. It is an advanced technology that allows the individual to move into a virtual environment and focus his attention on other thoughts to less consideration for pain and anxiety. In this study, VR glasses will be worn on the intervention group just before the procedure begins and patients will continue to wear their glasses until the procedure is completed.
  Arms: Intervention group

SUMMARY:
Coronary angiography (CAG) is a diagnostic method used as the gold standard in the diagnosis of coronary artery disease (CAD), which is increasingly prevalent in developed and developing countries and is one of the leading causes of morbidity and mortality in the world. Although coronary angiography is one of the best diagnostic methods of CAD, it can cause psychological problems such as stress, fear, anxiety in patients; It also causes physical problems such as bleeding, hematom and pain. Pharmacological and non-pharmacological methods are used by nurses to solve problems of patients, to ensure their relaxation and to improve their quality of life. With the development of technology, virtual reality (VR) glasses have been used to have fun at first, and later to provide pain management and to solve anxiety problems. VR glasses are an advanced technology that allows the patient to move into a virtual world and focus his attention on other thoughts, giving less attention to pain and anxiety. During literature search, no studies were found about the effect of using SG glasses on pain and anxiety during CAG. This research will be conducted to determine the effect of VR glasses used during CAG on pain, anxiety and hemodynamic parameters of patients who will experience coronary angiography for the first time.

DETAILED DESCRIPTION:
Although coronary angiography is widely used in the diagnosis and evaluation of CAD and heart valve diseases, it causes patients to experience intense stress, anxiety, pain and even fear of death. The main purpose of nurses before an interventional procedure is to increase the physiological and mental well-being of the patient and to help them adapt to the procedure. Various pharmacological and non-pharmacological methods are used to manage the psychological and physical problems of patients undergoing coronary angiography. Distraction is one of the non-pharmacological interventions commonly used during medical procedures. Virtual reality (VR) is a new method that can be used to distract and prepare patients for the procedure during medical procedures. It is thought to be more effective than traditional methods. Virtual reality is a computer-generated environment in which three-dimensional interaction is possible. It projects a wide field of view in front of the user's eye through advanced head-worn screens (glasses). It is an advanced technology that allows the individual to move into a virtual environment and focus his attention on other thoughts to less consideration for pain and anxiety.

This study is a randomized controlled study to determine the effectiveness of virtual reality glasses on pain, anxiety and hemodynamic parameters during coronary angiography.The universe of the study will be the individuals who will have a coronary angiography in the Angiography Laboratory of the Department of Cardiology, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital. On the other hand, the sample of the study will consist of patients who meet the inclusion criteria within the time the study is planned. Power analysis was performed using the G * Power (v3.1.7) program to determine the number of samples. It was decided that there should be at least 64 people in the groups. Participants in the study will be randomly divided into two groups as intervention and control groups. Before the procedure, patients will be informed about the purpose of the study, and written and verbal informed consent will be obtained from the patients. Patients in both groups will be asked to fill in the Personal Information Form before the procedure, and their pain levels will be evaluated with the Visual Analogue Scale (VAS), and their anxiety levels will be evaluated with the State-Trait Anxiety Inventory I (STAI-I). Immediately after the procedure, the pain levels of the patients with VAS and their anxiety levels will be evaluated with STAI-I. Virtual reality glasses will be worn on the intervention group just before the procedure starts and patients will continue to wear VR glasses until the procedure is completed. In patients selected as the control group, the same evaluations will be made at the same time interval. SPSS 22.0 (Statistical Package of Social Sciences) package program will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* To experience coronary angiography for the first time
* Not having contraindications for coronary angiography
* Not having visual and hearing impairment
* To be orientation to place, time and person
* Not having mental deficiency
* Not being addicted to alcohol and drugs
* Not being diagnosed with a psychiatric illness
* Having agreed to participate in research

Exclusion Criteria:

* Having undergone a treatment procedure (stent, balloon, etc.) during coronary angiography
* Having had a radial coronary angiography
* Not wanting to participate in the study
* Have used any painkillers at least 5 hours before coronary angiography
* Making coronary angiography decision under emergency conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change on pain intensity as measured by Visual Analog Scale | 'just before procedure and 30 minutes after procedure
  The average score change on pain intensity as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure pain intensity. The scale is a measuring tool with length of 0-10 cm. High scores on the scale indicate that pain intensity is high.

SECONDARY OUTCOMES:
Score change on anxiety level as measured by State-Trait Anxiety Inventory | just before procedure and 30 minutes after procedure
  The average score change on anxiety level as measured by State-Trait Anxiety Inventory. This scale in used to measure anxiety. The scores on the scale ranges from 20 to 80. The high scores on the scale indicate that anxiety is high.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ermis, Study Chair — Saglik Bilimleri University
Locations (1):
- University of Sağlık Bilimleri, Istanbul, Turkey (Türkiye)